CLINICAL TRIAL: NCT04874571
Title: Effect of Muscle Energy Technique on Clinical and Functional Levels in Chronic
Brief Title: Effect of Muscle Energy Technique on Clinical and Functional Levels in Chronic Obstructive Pulmonary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Serpil Mıhçıoğlu, Research assistant, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSerpil
Record Dates: First submitted 2021-05-03; First posted 2021-05-05 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Copd
Keywords: muscle energy technique; pulmonary disease; pain; home exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique group (Experimental): In the first group, according to Lewit's post-isometric relaxation (Muscle energy technique) method, scalene (anterior / medius / posterior), levator scapula, sternocleidomastoid, trapezius, pectoral muscles, serratus anterior and latismus dorsi muscles are set 3 days a week ( Each set includes three repetitions) The treatment will be applied for 4 weeks. The hypertonic muscle will be taken to the first point that resists movement without straining. The patient will be asked to perform an isometric contraction for 7 seconds, corresponding to 20% of the maximum isometric contraction force where the restriction is felt. After the application, the patient will be asked to exhale and relax completely. 30 seconds will be waited for each stretching and then the neck will be taken back to the barrier point and three repetitions per session will be performed.
  Interventions: Other: Muscle Energy Technique group
- Home Exercise (Other): The individuals in the second group will be asked to do the home exercise program shown to them for 4 weeks, 3 days a week. Individuals included in this group will be given a program that includes stretching and posture exercises for the same muscle groups. Individuals in the control group will be called weekly during the 4-week period. Before, after, and 6 weeks after the study, re-evaluation parameters will be applied to all individuals included in the study.
  Interventions: Other: Muscle Energy Technique group

INTERVENTIONS:
Other: Muscle Energy Technique group — In addition to the home exercise program of 12 sessions for 4 weeks, 3 days a week, muscle energy technique will be applied to the individuals in the MET(Musculer Energy Technique) group.

SUMMARY:
The primary aim of this study is to examine the effect on pain characteristics by applying muscle energy technique to patients with moderate chronic obstructive pulmonary disease.Secondary aim, clinical status of muscle energy technique in moderate chronic obstructive pulmonary patients: assessment of dyspnea and functional levels: kinesiophobia, muscle strength and endurance of neck muscles, hand grip strength, functional capacity, daily living activity, exercise habits, exercise efficiency, self-confidence, posture and to examine its effects on quality of life.

52 volunteer participants, 35 and 65 years old, diagnosed with moderate COPD, will be divided into muscle energy technique group (MET) (n = 26) and control group (CG) (n = 26) using randomization (minimization) method.

Individuals in the KET group will be applied muscle energy technique to certain muscles (Scalene(anterior-medius-posterior),Levator scapula,Sternocloidomastoideus, Upper trapezius, Pectoral muscles, Serratus anterior, Latissimus dorsi muscles) 3 days a week for 4 weeks and home exercise program applications will be requested. Individuals to be included in the study as a control group will be asked to apply home exercise programs 3 days a week for 4 weeks. All individuals included in the study will be re-evaluated parameters before, after and 6 weeks after the study.

In our study, the sociodemeographic information of the individuals who signed the voluntary consent form will be recorded. Pain Intensity Visual Analogue Scale (VAS), pain screening and evaluation of clinical features Brief Pain Inventory, pressure pain threshold of trapezoidal muscle and cervical paravertebral muscles with algometer, assessment of dyspnea with Medical Research Council (MRC) Dyspnea Scale, Fear of re-injury due to movement and activity Using the Tampa Kinesophobia Scale (TKS), measurement of muscle strength of neck muscles Digital Hand-Held Dynamometer (HHD), evaluation of neck muscles endurance with body weight and sandbag measurement of hand grip strength Hand Grip dynamometer, with the six-minute walking test of functional capacity, daily life activity with the Glittre GYA test, effectiveness of exercise Exercise wounds and barriers scale, Postural analysis with Newyork Posture Scale, health-related quality of life the St. George's Respiratory Questionnaire (SGRQ), general health-related quality of life Short Form SF-36 questionnaire will be evaluated using.

DETAILED DESCRIPTION:
DATA COLLECTION TOOLS AND FEATURES:

1. Demographic Information Age, gender, height, weight, body mass index (BMI), profession, dominant side, educational status, history, family history, smoking and alcohol consumption, medications used, pain, pain Exercise behavior, injury mechanism (previous sports injuries, accidents) and location and duration of symptoms, COPD exacerbation history, exercise effectiveness and self-confidence will be recorded.
2. Pain Assessment 2.1. Visual Analogue Scale (GAS) The severity of pain during rest, activity and night time will be evaluated by VAS.

   2.2. Brief Pain Inventory (BPI) The short pain questionnaire (BPI) is a multi-dimensional pain assessment scale that has been validated in Turkish and is easy to apply. This scale will evaluate the presence of pain, severity, character, treatments, responses to this treatment, general activity, and social-emotional effects on the basis of the last week of the patients. The severity of each item will be graded from 0 (no obstacle) to 10 (obstruction). It consists of 32 questions in total.

   2.3. Evaluation of Pressure Pain Thresholds The pressure pain threshold will be evaluated with a digital algometer, which is an objective assessment method. The pain thresholds of the upper trapezoidal and cervical paravertebral muscles will be evaluated using the QST Pressure Pain Threshold branded algometer device. Trapezius muscle tenderness will be evaluated from 3 points: medial of acromion, body of muscle and 7th vertebra level. Cervical paravertebral muscle sensitivity will be evaluated from 3 points: C1 level, between C3 and C4, and C7. All measurements will be evaluated by the same physiotherapist with the same algometer.
3. Assessment of Fear of Movement The Tampa Kinesophobia Scale (TKS) is a 17-question scale developed to measure fear of re-injury due to movement and activity. This scale includes fear, avoidance and re-injury parameters in work-related activities.
4. Evaluation of Cervical Region Muscle Strength 4.1.Muscle strength measurement of the cervical flexor muscles will be evaluated in the supine position in the head and neck neutral position, the arms at the side of the trunk, and the knees in the extension position. With the help of Velcro, the body will be fixed to the bed over the spina iliaca anterior superior and sternum. Contraction will be requested from individuals against Hand-held Dynamometer(HHD) placed on the frontal bone.

4.2. Measurement of the strength of the cervical extensor muscles will be made in the prone position, with the head and neck in neutral, and the arms in a free position next to the body. With the help of Velcro, the measurement will be made by fixing the body to the bed over the spina iliaca posterior superior and T3 vertebra. Contraction will be desired by placing the HHD in the occipital area.

4.3. While the neck lateral flexor and rotator muscle strengths are measured, the patient will be seated in a chair with back support, with his hands tied to his body. With the head in a neutral position, the dynamometer for rotators will be placed on the external auditory canal, in the center of rotation.

4.4. For lateral flexors, the dynamometer will be placed on the head over the ear in a position that prevents movement. The patient will be told the movement to do with his head in neutral, and measurements will be made in a way that does not allow the patient's head to move.

5 seconds for each test. During the contraction will be requested and the tests will be repeated 3 times and the best value will be recorded in kilograms (kg). There will be a 15-second rest break between repetitions and a 2-minute rest break between movements.

5. EVALUATION OF THE CERVICAL AREA ENDURANCE 5.1. Endurance Evaluation of Cervical Region Flexor Muscles In evaluating the neck flexors muscles endurance, individuals will be asked to lie on their back with the hands on the side of the body and the knees in a 90-degree position. The hand of the physiotherapist will be placed under the head of the individuals and they will be asked to gently press the chin backwards with two fingers (after the chin is in the tuck position) and lift the head approximately 2.5 cm from the bed, to protect this position without disturbing it. The time in which the individual can maintain this position will be recorded in seconds. The test will be terminated when he is unable to maintain the position due to any pain or fatigue or if the physiotherapist touches his hand.

5.2. Endurance Evaluation of Cervical Extensor Muscles In order to evaluate the endurance of the deep and superficial extensor muscles of the neck, the patients will be asked to hang down from the bed in the prone position, arms by the trunk, head to the thoracic 6 vertebra level. While all individuals are in neutral position, 4 kg weight for men and 2 kg for women will be fixed with the help of a velcro from the occiput level of the head and the test will start, motivating words will not be used during the test. Individuals will be asked to maintain this position and the time will be recorded in seconds. The test will be terminated if there is a 5 degree change in the head position 6. Assessment of Hand Grip Strength The procedure recommended by the American Association of Hand Therapists (ASHT) for hand grip strength measurement will be applied.

7. Assessment of Shortness of Breath Modified Medical Research Council (MMRC) Dyspnea Scale will be used to evaluate the perception of dyspnea.

8. Assessment of Functional Capacity The Six Minute Walking Test (6 MWT), which is considered a gold standard in individuals with COPD, is an easy test that evaluates the distance that individuals walk for six minutes. 6 DYT will be conducted according to the American Thoracic Society (ATS) rules. Standardized 6 DYT will be applied according to ATS.

9.Glittre Daily Living Activity Assessment The test begins with the person sitting in a chair. During the test, a backpack weighing 2.5 kg for women and 5 kg for men is attached. Standing up from the chair, he walks 5 m and passes a 2-step ladder placed in the middle with a width of 17 cm and a depth of 27 cm, and walks another 5 m to a 2-shelf setup that is individually adjusted according to the shoulder and waist height of the individual. Three bottles, each weighing 1 kg, placed on the upper rack must be transported one by one to the lower rack, to the floor, to the lower rack, and finally to the upper rack. Then the participants pass the 2-step stairs, return to the original chair, sit down and immediately rise again and begin the next round. They will be allowed to rest if necessary, but the stopwatch will continue to run during this time. Individuals are asked to complete 5 rounds quickly, and the time is recorded in minutes after 5 rounds. Heart rate, blood pressure, saturation, fatigue and shortness of breath are evaluated at the beginning and end of the test.

10. Posture Evaluation The postures of the subjects participating in the study will be evaluated with the "New York Posture Assessment Method (NYPDY)". In this evaluation system, posture changes that may occur in 13 different parts of the body will be followed and scored.

11.Exercise Habits Exercise benefit / disability scale was developed by Sechrist, Walker, and Pender to determine exercise benefit and disability perceptions of individuals participating in exercise.The scale consists of 43 items in total.

12. Quality of Life 12.1. St. George Respiratory Questionnaire Among the tests measuring the quality of life related to health, especially St. St. George's Respiratory Questionnaire (SGRQ) is a specific test for respiratory diseases. SGRQ questions 50 items in the patient, distributed over three areas = Symptoms (8 items), activities (16 items), effects of the disease (26 items).

12.2. Short Form 36 (Short Form 36 / SF 36) Short Form 36 is a valid health questionnaire with 36 questions providing information about functional health and well-being. It provides valid and reliable information about psychometric-based mental and physical health, which can be filled in as short as five to 10 minutes.

Treatment protocol:

All individuals will be divided into 2 groups by randomization method. In the first group, according to Lewit's post-isometric relaxation (KET) method, scalene (anterior / medius / posterior), levator scapula, sternocleidomastoid, trapezius, pectoral muscles, serratus anterior and latismus dorsi muscles are set 3 days a week ( Each set includes three repetitions) The treatment will be applied for 4 weeks. The hypertonic muscle will be taken to the first point that resists movement without straining. The patient will be asked to perform an isometric contraction for 7 seconds, corresponding to 20% of the maximum isometric contraction force where the restriction is felt. After the application, the patient will be asked to exhale and relax completely. 30 seconds will be waited for each stretching and then the neck will be taken back to the barrier point and three repetitions per session will be performed.

The individuals in the second group will be asked to do the home exercise program shown to them for 4 weeks, 3 days a week. Individuals included in this group will be given a program that includes stretching and posture exercises for the same muscle groups. Individuals in the control group will be called weekly during the 4-week period. Before, after, and 6 weeks after the study, re-evaluation parameters will be applied to all individuals included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 35-65,
* Moderate COPD diagnosed according to Gold criteria by a chest diseases specialist,
* Neck pain longer than 3 months
* Those who are not diagnosed with fibromyalgia will be included in the study.

Exclusion Criteria:

* COPD exacerbation period,
* Those with disc herniation, fracture, etc. musculoskeletal problems in the cervical and thoracic region
* Undergoing cervical surgery,
* Having problems preventing him from exercising,
* Those with uncontrolled diabetes, hypertension and coronary artery disease,
* Individuals who received physiotherapy due to neck pain in the last 3 months will not be included in the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Pain thresold | change from baseline at 4 weeks and 6 weeks after the intervention
  This is measured by using digital pressure algometry.

SECONDARY OUTCOMES:
Severity of pain | change from baseline at 4 weeks and 6 weeks after the intervention
  severity of pain is measured by Visual analogue scale. This is a scale including scores from 0 to 10. Zero means no pain and 10 means very severe pain and patients are asked to grade their pain on this scale for three times of the day as resting times, activity times and evening times.
Multidimensional pain assessment | change from baseline at 4 weeks and 6 weeks after the intervention
  The short pain questionnaire (BPI) is a multi-dimensional pain assessment scale that has been validated in Turkish and is easy to apply. This scale will evaluate the presence of pain, severity, character, treatments, responses to this treatment, general activity, and social-emotional effects on the basis of the last week of the patients. The severity of each item will be graded from 0 (no obstacle) to 10 (obstruction). It consists of 32 questions in total. The first 9 questions question the demographic characteristics of the patient, the presence of a previous operation and the pain before the illness.
Assessment of Fear of Movement | change from baseline at 4 weeks and 6 weeks after the intervention
  The Tampa Kinesophobia Scale (TKS) is a 17-question scale developed to measure fear of re-injury due to movement and activity. This scale includes fear, avoidance and re-injury parameters in work-related activities. Likert scoring of 4 points (1 = Strongly disagree-4 = Strongly agree) is used in TKS. The total score is between 17-68. The higher his score as a result of the scale indicates that his kinesiophobia is also high.
Evaluation of Cervical Region Muscle Strength | change from baseline at 4 weeks and 6 weeks after the intervention
  Measurement of the muscle strength of the neck muscles will be done using a Digital Hand-held Dynamometer (HHD). Muscular strengths of cervical flexors, extensors, lateral flexors and rotators of both sides of all individuals will be evaluated.
Endurance Evaluation of Cervical Region Flexor Muscles | change from baseline at 4 weeks and 6 weeks after the intervention
  In evaluating the neck flexors muscles endurance, individuals will be asked to lie on their back with the hands on the side of the body and the knees in a 90-degree position. The hand of the physiotherapist will be placed under the head of the individuals and they will be asked to gently press the chin backwards with two fingers (after the chin is in the tuck position) and lift the head approximately 2.5 cm from the bed, to protect this position without disturbing it. The time in which the individual can maintain this position will be recorded in seconds.
Endurance Evaluation of Cervical Extensor Muscles | change from baseline at 4 weeks and 6 weeks after the intervention
  In order to evaluate the endurance of the deep and superficial extensor muscles of the neck, the patients will be asked to hang down from the bed in the prone position, arms by the trunk, head to the thoracic 6 vertebra level. While all individuals are in neutral position, 4 kg weight for men and 2 kg for women will be fixed with the help of a velcro from the occiput level of the head and the test will start, motivating words will not be used during the test. Individuals will be asked to maintain this position and the time will be recorded in seconds.
Assessment of Hand Grip Strength | change from baseline at 4 weeks and 6 weeks after the intervention
  The procedure recommended by the American Association of Hand Therapists (ASHT) for hand grip strength measurement will be applied. They suggested that individuals should be measured in a sitting position on a chair with back support without armrests, shoulder adduction, elbow 90 ° flexion, forearm in neutral position, wrist 15 to 30 ° dorsiflexion and 0-15 ° ulnar lead. To prevent the effect of gravity on maximum force, the physiotherapist will support the dynamometer from below. The measurements will be repeated 3 times for the right and left hand and averaged. There will be a 30-second rest break between each measurement to prevent fatigue.
Assessment of Shortness of Breath | change from baseline at 4 weeks and 6 weeks after the intervention
  Modified Medical Research Council (MMRC) Dyspnea Scale will be used to evaluate the perception of dyspnea. The MMRC Dyspnea Scale is a 0-4 point scale in which patients choose the statement that best describes their dyspnea level among 5 statements about dyspnea.
Assessment of Functional Capacity | change from baseline at 4 weeks and 6 weeks after the intervention
  The Six Minute Walking Test (6 MWT), which is considered a gold standard in individuals with COPD, is an easy test that evaluates the distance that individuals walk for six minutes. 6 DYT will be conducted according to the American Thoracic Society (ATS) rules.
Glittre Daily Living Activity Assessment | change from baseline at 4 weeks and 6 weeks after the intervention
  The test begins with the person sitting in a chair. During the test, a backpack weighing 2.5 kg for women and 5 kg for men is attached. Standing up from the chair, he walks 5 m and passes a 2-step ladder placed in the middle with a width of 17 cm and a depth of 27 cm, and walks another 5 m to a 2-shelf setup that is individually adjusted according to the shoulder and waist height of the individual. Three bottles, each weighing 1 kg, placed on the upper rack must be transported one by one to the lower rack, to the floor, to the lower rack, and finally to the upper rack. Then the participants pass the 2-step stairs, return to the original chair, sit down and immediately rise again and begin the next round.
Posture Evaluation | change from baseline at 4 weeks and 6 weeks after the intervention
  The postures of the subjects participating in the study will be evaluated with the "New York Posture Assessment Method (NYPDY)". In this evaluation system, posture changes that may occur in 13 different parts of the body will be followed and scored.
Exercise Habits | change from baseline at 4 weeks and 6 weeks after the intervention
  Exercise benefit / disability scale was developed by Sechrist, Walker, and Pender to determine exercise benefit and disability perceptions of individuals participating in exercise.The scale consists of 43 items in total.
Measuring the quality of life related to health | change from baseline at 4 weeks and 6 weeks after the intervention
  Among the tests measuring the quality of life related to health, especially St. St. George's Respiratory Questionnaire (SGRQ) is a specific test for respiratory diseases.
İnformation about functional health and well-being | change from baseline at 4 weeks and 6 weeks after the intervention
  Short Form 36 is a valid health questionnaire with 36 questions providing information about functional health and well-being. It provides valid and reliable information about psychometric-based mental and physical health, which can be filled in as short as five to 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Mehtap MALKOÇ, Prof.Dr., Study Director — Eastern Mediterranean University
Locations (1):
- Serpil MIHÇIOĞLU, Famagusta, Cyprus

REFERENCES:
- [Derived] Mihcioglu S, Malkoc M. Effect of muscle energy technique on pain, importance of physical activity, self-confidence, and posture in COPD patients with chronic neck pain: An experimental randomized controlled study. Medicine (Baltimore). 2025 Jun 20;104(25):e42849. doi: 10.1097/MD.0000000000042849. PMID 40550078
- [Derived] Mihcioglu S, Malkoc M. The effect of muscle energy technique on pain, kinesiophobia, and quality of life in patients with COPD with chronic pain. Sci Rep. 2025 Jan 31;15(1):3884. doi: 10.1038/s41598-025-88304-w. PMID 39890971